CLINICAL TRIAL: NCT03261648
Title: Anxiety of Patient and His Partner During Admission to Emergency Department
Acronym: ANXURG
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17-0033; 2017-A00511-52 (Other: ID-RCB)
Record Dates: First submitted 2017-07-27; First posted 2017-08-25 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Anxiety; Emergencies
MeSH Terms: conditions — Anxiety Disorders; Emergencies | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hospitalized patient: 100 patients will completed the 'State-Trait-Anxiety Inventory (Forme Y) questionnaire Patients will evaluated here pain answering to a pain level scale
  Interventions: Other: State-Trait-Anxiety Inventory (Forme Y) questionnaire; Other: pain level scale
- partner of the hospitalized patient: 100 partners will completed the State-Trait-Anxiety Inventory (Forme Y) questionnaire
  Interventions: Other: State-Trait-Anxiety Inventory (Forme Y) questionnaire

INTERVENTIONS:
Other: State-Trait-Anxiety Inventory (Forme Y) questionnaire — after admission in the emergency department, patient and his partner will completed STAI Y questionnaire.
Other: pain level scale — as usual caregiver will ask to the patient to evaluated his pain level with a scale of one to ten
  Groups: hospitalized patient

SUMMARY:
Evaluate and compare the impact of partner's stress in the pain of the patient admitted in the emergency department

DETAILED DESCRIPTION:
Admission to an emergency department is a major source of anxiety for the patient. Anxiety plays not only a role in its emotional state but can also have consequences on the taking care of the patient and especially on the analgesic procedure.

Since pain is one of the first causes of emergency admission, patient anxiety should not be overlooked. In the emergency department, patient consults frequently, with his partner . Anxiety can also affect the partner, which may affect the patient. No studies have yet demonstrated this correlation.

This study will evaluate, the anxiety of both parties and show the presence or not of an influence of the partner's anxiety on the patient using a standardized questionnaire, the State-Trait Anxiety Inventory- form Y (STAI-Y).

ELIGIBILITY:
Inclusion Criteria:

* Admission to emergency department accompanied by his partner (lives in concubinage with the patient)
* Nurse patient's classification score up or equal to 3, 4 or 5
* Oral consent given to the inclusion by the patient and the partner
* Patient and partner Francophone or with a good understanding of French

Exclusion Criteria:

* Patient under a system of legal protection
* Non-Communicating Patient and partner
* Patient and partner unable to write
* Refusal of patient or partner
* Admission of the patient with shock treatment corresponding to the nurse patient's classification score 1 and 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people admited in the emergency department and his partner
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Compare the anxiety of the patient with that of his partner | day 1
  The anxiety will be evaluated by the State-Trait-Anxiety Inventory (Forme Y) questionnaire

SECONDARY OUTCOMES:
Study the link between the patient's and his partner's anxiety | day 1
  A corelation will be do between the score obtained by the patient and the score obtained by the partner at the STAI-Y questionnaire
Evaluate the link between the patient's anxiety and the patient's pain | day 1
  The patient's pain will be evaluated orally asking to him to use a scale pain to 0 of 10

CONTACTS AND LOCATIONS:
Overall Officials: Vincent BOUNES, MD, Principal Investigator — University Hospital of Toulouse, Toulouse, France
Locations (1):
- University Hospital of Toulouse, Toulouse, France